CLINICAL TRIAL: NCT07342894
Title: Effect of Timing of Hemovac Drain Removal on Early Outcomes After Total Knee Arthroplasty
Brief Title: Effect of Hemovac Drain Removal on Early Outcomes After Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Şahan Güven, Medical Doctor, specialist, Ankara City Hospital Bilkent
Other Study IDs: TABED2-25-1015_TKA_DRAIN
Record Dates: First submitted 2025-12-22; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Knee Osteoarthritis; Total Knee Arthroplasty
Keywords: Knee Osteoarthritis; Total Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early Drain Removal (Goup 1): Patients whose Hemovac drain is removed before the first postoperative rehabilitation session as part of routine clinical practice.
- Late Drain Removal (Group 2): Patients whose Hemovac drain is removed after completion of the first postoperative rehabilitation session as part of routine clinical practice.

SUMMARY:
This study aims to evaluate whether the timing of Hemovac drain removal affects early clinical outcomes after primary total knee arthroplasty (TKA). Hemovac drains are commonly used after TKA to reduce postoperative bleeding and swelling; however, the optimal timing for drain removal remains controversial.

In this prospective observational cohort study, patients undergoing primary TKA for knee osteoarthritis will be divided into two groups according to routine clinical practice: those whose drain is removed before the first postoperative rehabilitation session and those whose drain is removed after the first rehabilitation session.

The primary outcomes include the rate of postoperative hemarthrosis, early postoperative complications, and length of hospital stay. Secondary outcomes include postoperative pain levels and functional outcomes. The results of this study may help optimize postoperative management strategies following total knee arthroplasty.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is a widely performed surgical procedure for the treatment of advanced knee osteoarthritis. Postoperative management often includes the use of closed suction drains, such as Hemovac systems, to reduce hematoma formation and wound complications. However, the necessity and optimal timing of drain removal remain subjects of debate.

This prospective observational cohort study is designed to compare early clinical outcomes associated with two different timings of Hemovac drain removal following primary TKA. Patients who undergo primary TKA at a single tertiary care center will be enrolled prospectively. According to routine postoperative practice, patients will be allocated into two groups: drain removal before the first postoperative rehabilitation session or drain removal after completion of the first rehabilitation session.

All patients will receive standardized surgical techniques, anesthesia protocols, postoperative care, and rehabilitation programs. Data will be collected prospectively. Primary outcomes include postoperative hemarthrosis, early postoperative complications, and length of hospital stay. Secondary outcomes include postoperative pain intensity and functional outcome measures.

This study aims to provide evidence to guide clinical decision-making regarding postoperative drain management in patients undergoing total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Diagnosis of knee osteoarthritis
* Undergoing primary total knee arthroplasty
* Provided written informed consent to participate in the study

Exclusion Criteria:

* Revision total knee arthroplasty
* History of inflammatory arthritis
* Known bleeding disorders or coagulopathy
* Active infection or periprosthetic joint infection
* Incomplete clinical data or loss to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients diagnosed with knee osteoarthritis who underwent primary total knee arthroplasty at a single tertiary care center. All participants were treated according to standardized surgical and postoperative care protocols and were followed prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Postoperative Drain Output | Postoperative days 0-3
  Total postoperative Hemovac drain output measured in milliliters following primary total knee arthroplasty.

SECONDARY OUTCOMES:
Length of Hospital Stay | Postoperative days 0-discharge
  Duration of postoperative hospital stay measured in days.
Postoperative Hemoglobin Change | Postoperative first 24-48 hours
  Change in hemoglobin level from preoperative baseline to postoperative measurement.
Knee Society Score (KSS) | Postoperative 1 month
  Functional outcome assessed using the Knee Society Score.
Postoperative Pain Intensity | Postoperative 1 month
  Pain intensity assessed using the Visual Analog Scale (VAS).

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No